CLINICAL TRIAL: NCT02694237
Title: The Age of OrthoInfo: A Randomized Controlled Trial Evaluating Patient Comprehension of Informed Consent in a Private Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Nkemakolam Egekeze, UMKC Orthopaedic Research Fellow, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoInfo
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Models, Biological; Memory and Learning Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Verbal (Active Comparator): This group will only receive a verbal discussion based on the same script used for all three groups. This is the control group.
  Interventions: Behavioral: Verbal
- Verbal + Model (Active Comparator): This group will receive a verbal discussion aided with an anatomic model intervention that group participants will be able to touch throughout the discussion.
  Interventions: Behavioral: Model
- Verbal + Video (Active Comparator): This group will receive a verbal discussion aided with a knee anatomy video intervention that will be played on silent an orated by an interviewer.
  Interventions: Behavioral: Knee Anatomy Video

INTERVENTIONS:
Behavioral: Model — Each participant will receive an informed consent discussion with the aid of an anatomic knee model.
  Arms: Verbal + Model
Behavioral: Knee Anatomy Video — Each participant will hear a scripted informed consent discussion while they watch a knee anatomy video orated by an interviewer.
  Arms: Verbal + Video
Behavioral: Verbal — Each participant will receive a verbal informed consent discussion without a visual aid.
  Arms: Verbal

SUMMARY:
The aim of the study is determine which method of informed consent improves comprehension in college educated patients in a private practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis patients over the age of 18 with a college education deemed appropriate for medical management with a knee injection.

Exclusion Criteria:

* Patients without the capacity to provide consent
* Patients with a visual, auditory, psychological or tactile impairment requiring the assistance of another person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The Nkem Test | baseline
  This knowledge based questionnaire assesses patient comprehension of an informed consent discussion. The score of the test is known as "The Nkem Score".

CONTACTS AND LOCATIONS:
Overall Officials: Nkem Egekeze, MD, Principal Investigator — UMKC Department of Orthopaedic Surgery; Karen Williams, PhD, Study Director — UMKC Department of Health Insight and Research; Luv Singh, MD, Study Director — UMKC Department of Orthopaedic Surgery; Dan Gurba, MD, Study Director — Dickson-Diveley Orthopaedic Clinic; Charles Rhoades, MD, Study Director — UMKC Department of Orthopaedic Surgery; Mark Bernhardt, MD, Study Chair — UMKC Dept of Orthopaedic Surgery
Locations (1):
- Truman Medical Center and Dickson-Diveley Orthopaedic Clinic, Kansas City, Missouri, United States